CLINICAL TRIAL: NCT04056637
Title: Choice of Modality of Follow up for Medication Abortion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Impacted Service Delivery and Research Infrastructure
Sponsor: Stanford University (Other)
Collaborators: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 52312
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Abortion in First Trimester
Keywords: MLPT; multi-level pregnancy test; medication abortion; first trimester abortion; abortion follow-up

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Standard of Care (No Intervention): Participants will be asked to complete follow-up in clinic 1-2 weeks following mifepristone administration for an ultrasound and consultation with a provider.
- Group 2: Flexible Follow-Up (Experimental): Participants will be offered three follow-up options, including: 1) follow-up in clinic 1-2 weeks following mifepristone administration for an ultrasound and consultation with a provider; 2) repeat serum beta-hCG testing; 3) repeat multi-level pregnancy test strategy
  Interventions: Other: Choice of follow-up option; Device: Multi-level pregnancy test

INTERVENTIONS:
Other: Choice of follow-up option — Participant will be given the opportunity to choose from 3 follow-up options.
  Arms: Group 2: Flexible Follow-Up
Device: Multi-level pregnancy test — The Multi-level pregnancy test (MLPT) strategy involves the use of the MLPT to estimate a pregnant person's baseline hCG range prior to beginning their abortion (i.e. prior to mifepristone administration). A follow-up test is then administered one week later to again estimate the woman's hCG range. A decline in hCG range reliably signifies absence of an ongoing pregnancy. Among clients ≤63 days' LMP at initiation of treatment, this strategy has shown to be highly effective: 100% of clients (n=1487/1487) with a decline in hCG range did not have an ongoing pregnancy and 100% of clients (n=21/21) with an ongoing pregnancy showed steady or increase in hCG range on their follow-up MLPT.
  Other Names: dBest
  Arms: Group 2: Flexible Follow-Up

SUMMARY:
This study will assess the impact of providing medication abortion-seeking clients a choice for follow-up in practice. Clients presenting at or less than 63 days pregnant (based on last menstrual period) at the study site for first trimester medication abortion will be invited to participate. We hypothesize that providing clients with flexible follow-up options will improve follow-up rates.

This study is not to assess efficacy or safety of follow-up methods--that has been well established in practice and research. This is to assess choice of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for medication abortion <63 days gestational age
* In general good health
* English or Spanish speaking competency
* Willing and able to sign consent forms

Exclusion Criteria:

* Clients less than 18 years of age.
* Any client not meeting the inclusion criteria listed above will be excluded from participating in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Percent follow-up after medication abortion by group | 5-14 days following mifepristone administration
  To compare rates of follow-up among clients who are instructed to come back to the clinic for in-person ultrasound medication abortion follow-up to clients who are given options for follow-up, including in-person ultrasound, repeat serum beta-hCG and MLPT

SECONDARY OUTCOMES:
Percent follow-up after medication abortion by follow-up type | 5-14 days following mifepristone administration
  To compare the overall proportion of follow-up completion among clients choosing their preferred method of follow-up (in-person ultrasound, repeat serum beta-hCG, MLPT strategy) (study period) to clients given only the option for in-person follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared.